CLINICAL TRIAL: NCT03210363
Title: Sero-epidemiology of Priority Arboviruses in French Guiana
Acronym: EPI-ARBO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Pasteur (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2016-073
Record Dates: First submitted 2017-06-16; First posted 2017-07-06 (Actual); Last update posted 2020-09-14 (Actual); Status verified 2020-09

CONDITIONS: Arbovirus Infections
MeSH Terms: conditions — Arbovirus Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Guiana population (Experimental): Human Biological samples from Guiana population :
  Two serum tubes of blood will be collected
  Interventions: Other: Human Biological samples

INTERVENTIONS:
Other: Human Biological samples — Blood sample

SUMMARY:
Dengue is an important public health problem despite the efforts of local health authorities to mitigate the impact of epidemics and the epidemiology of dengue evolved from an endemo-epidemic to a hyper-endemic state. In late 2013, the first local transmission of chikungunya virus in the Americas was identified in Caribbean countries and territories including French Guiana. Rapidly, more than 16,000 suspected local Health authorities had reported cases. In May 2015, the Pan American Health Organization (PAHO) issued an alert regarding the first confirmed Zika virus infections in Brazil. The emergence of Zika virus in South America led to a rapid spread throughout South and Central America, reaching French Guiana in December 2015. With the increasing frequency of epidemics related to arbovirus and the resulting health, social, and economic impacts of dengue, the surveillance of arbovirus have become social, political, and public health challenges that require specific and non-available immune status information.

DETAILED DESCRIPTION:
French Guiana is a 250,000 inhabitant's French overseas department located in South America, the epidemiology of arboviruses has recently evolved and marked by important outbreaks.

Dengue remains an important public health problem despite the efforts of local health authorities to mitigate the impact of epidemics and the epidemiology of dengue evolved from an endemo-epidemic to a hyper-endemic state. In late 2013, the first local transmission of chikungunya virus in the Americas was identified in Caribbean countries and territories including French Guiana. Rapidly, more than 16,000 suspected local Health authorities had reported cases. In May 2015, the Pan American Health Organization (PAHO) issued an alert regarding the first confirmed Zika virus infections in Brazil. The emergence of Zika virus in South America led to a rapid spread throughout South and Central America, reaching French Guiana in December 2015. With the increasing frequency of epidemics related to arbovirus and the resulting health, social, and economic impacts of dengue, the surveillance of arbovirus have become social, political, and public health challenges that require specific and non-available immune status information.

ELIGIBILITY:
Inclusion Criteria:

* Guiana resident for at least 6 months and present during the entire study period
* Age between 2 and 75 years old

Exclusion Criteria:

* Subject under guardianship or deprived of liberty by judicial decision
* Subject with any pathology or health problem not compatible with blood sampling

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 2697 (Actual)
Dates: Start 2017-06-09 (Actual); Primary Completion 2017-11-21 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Dengue, chikungunya, zika Antibodies detection by multiplex serologic tests | 2 years
  Description of the virological status of individuals by Mutiplex detection of antibodies directed against dengue, chikungunya and zika arboviruses.

SECONDARY OUTCOMES:
Seroprevalence by area and age | 2 years
  Estimatation of the frequency of Dengue, Chikungunya and zika infections among the general population of French Guiana by geographical area and by age class

OTHER OUTCOMES:
Dengue infections proportion | 2 years
  Proportion of dengue primary and multiple infections in Guiana population.

CONTACTS AND LOCATIONS:
Overall Officials: Claude Flamand, Principal Investigator — Institut Pasteur de la Guyane
Locations (1):
- Institut Pasteur de la Guyane, Cayenne, France

IPD SHARING:
Plan to Share IPD: No